CLINICAL TRIAL: NCT03281161
Title: Sun Safe Workplaces: Assessment of Benefits and Costs of a Policy Intervention
Acronym: SSW2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Kaiser Foundation Research Institute (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01CA187191-02 (NIH); 5R01CA187191-02 (NIH); 0284 (Other: Klein Buendel, Inc.)
Record Dates: First submitted 2017-09-06; First posted 2017-09-13 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Skin Cancer
Keywords: skin cancer; prevention; worksite; policy; cost and effectiveness; implementation
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not aware of the condition in which their organization was enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sun Safe Workplaces Program (Experimental): A follow up to the previous study that promoted the adoption of occupational sun protection policies by the local government organization comprised of personal visits with senior managers to promote policy adoption, promotional materials for sun safety, and in-person training of outdoor workers by research staff over two years. The follow up program consists of an analysis of sun safe practices by employees and an economic evaluation of the SSW intervention completed 2 years after the initial intervention.
  Interventions: Behavioral: Sun Safe Workplaces Program
- Attention Control (Active Comparator): A follow up to the previous study that promoted occupational sun protection practices by employees in local government organizations through two mailings containing educational materials and presentations at state professional meetings by project staff. The follow up program consists of an analysis of sun safe practices by employees and an economic evaluation of SSW completed 2 years after the initial program contact.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Sun Safe Workplaces Program — A follow-up analysis of sun safe practices by employees and an economic evaluation of the SSW intervention was conducted with the work-sites who received occupational sun protection policy promotion materials in the prior trial. The analysis of sun safety practices of employees was done by preparing the protocols and measures for surveying employees and front-line supervisors by online and paper methods. The economic evaluation was a retrospective collection of cost information from the prior project ledgers and an in depth interview with the key contact manager at each work-site. No additional treatment was provided and the groups were evaluated based on their prior condition assignment.
  Arms: Sun Safe Workplaces Program
Behavioral: Attention Control — A follow-up analysis of sun safe practices by employees and an economic evaluation of the SSW intervention was conducted with the work-sites who received occupational sun protection practice promotion materials in the prior trial. The analysis of sun safety practices of employees was done by preparing the protocols and measures for surveying employees and front-line supervisors by online and paper methods. The economic evaluation was a retrospective collection of cost information from the prior project ledgers and an in depth interview with the key contact manager at each work-site. No additional treatment was provided and the groups were evaluated based on their prior condition assignment.
  Arms: Attention Control

SUMMARY:
Sun Safe Workplaces (SSW), a comprehensive occupational sun safety program, promoted education and policy to 98 cities, counties, and special districts in Colorado. In a two-year follow-up study, Klein Buendel, Inc. (KB) proposes to examine the effectiveness of SSW on employee sun protection practices by employers and return on investment in an economic evaluation of the cost of the SSW intervention. The results of this follow-up study will provide critical information on effective approaches to increasing sun protection across a wide range of employment sectors with outdoor workers.

DETAILED DESCRIPTION:
Workers in the United States spend large amounts of time on the job, making the workplace a key venue for preventive health programs. A workplace risk that has received limited attention is solar ultraviolet radiation (UVR). Unprotected exposure to solar UVR of outdoor workers can produce both an immediate acute harm (i.e., severe sunburn) and long-term skin damage that can elevate the risk of developing skin cancers. Preventing skin cancer is a priority due to its high prevalence; tendency to recur; association with other cancers; and lost productivity ($66.9 billion in losses were attributed to melanoma-related mortality from 1990-2008). Sun Safe Workplaces (SSW) is a comprehensive occupational sun safety education and policy intervention that was tested by Klein Buendel, Inc.'s (KB) research team in a randomized control trial with 98 cities, counties, and special districts in Colorado. Posttesting was completed in November 2013. The SSW intervention focused on three sectors in the organizations: public works, public safety, and parks and recreation. Half of the employers received the SSW intervention, with the remaining employers in the control condition receiving basic sun safety information. Preliminary analyses indicate that 80% of employers in the SSW intervention condition provided sun safety education to employees and 36% adopted formal sun protection policies. No control organizations reported policy adoption. KB will conduct a two-year follow-up study on the benefits of the SSW intervention (i.e., increasing employees' sun protection) and return on investment (ROI; benefits relative to intervention costs). Employee behavior was not assessed in the current SSW trial because it was uncertain whether the SSW intervention would result in uptake of education and policy and thus have the potential to influence their sun protection practices. The proposed two-year follow-up of the 98 organizations in the SSW trial will include: (1) surveys with employees (n=10,787) and front line supervisors (n=767) to assess employees' sun protection practices and workplace actions to support employee sun safety; (2) on-site observations of sun protection actions by the employers (e.g., posters, sunscreen, shade structures); and (3) tracking of the costs of implementing the SSW intervention and induced employer costs. The proposed analyses will compare the sun protection practices of employees a) between workplaces that received the SSW intervention and controls and b) among workplaces that provided education and adopted policy, provided education only, and control workplaces. Analyses will determine if the extent of sun protection actions by employers influences employees' sun safety practices. The economic evaluation will estimate the ROI (i.e., comparison of the estimated program benefits to combined cost elements). The proposed study is significant and innovative because it provides critical information applicable to a wide range of industrial sectors with outdoor workers on a workplace risk that has received scant attention. Determining the effectiveness and ROI of prevention programs is essential for national and local resource investment.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the prior Sun Safe Workplaces: A Campaign on Sun Protection Policies for Outdoor Workers.
* A local government organization with employees who worked outdoors in at least one of the following service areas: public works, public safety, and parks and recreation,
* Having a full time executive
* Having a population of at least 3000 residents
* Being employed at a participating local government organization as a manager or employee?
* Being employed at a participating local government organization in a job requiring outdoor work at least part of the time.

Exclusion Criteria:

* Organization had participated in the authors' previous occupational sun protection project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1990 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Survey of sun protection practices by employees. | 9 Months
  Quantitative research in the form of a posttest survey was conducted to examine the sun safety practices by employees among workplaces that received education but did not adopt written policies, those workplaces that received education and adopted written policies and those that were in the control group.safety practices by employees among workplaces that received education but did not adopt written policies.

SECONDARY OUTCOMES:
Observational checklist to review sun protections items within the workplace. | 9 months
  An observational visit checklist was used to review sun protection items within the environment to assess employer actions to improve worker sun safety in the SSW parent study project. This checklist accounted for program materials (posters, tip cards, brochures, policy tool box items) and other sun safety protective items such as sunscreen and portable and permanent shade provided by the workplace for employees.
In-depth manager interview to assess relationship of employer sun safety actions to employee sun safety. | 9 Months
  Analysis of the association of employer actions (education only vs. education plus policy) on sun safety with employee's sun protection practices.
In-depth manager survey to assess relationship of employer sun safety actions to employee sun safety. | 9 Months
  Analysis of the association of employer actions (education only vs. education plus policy) on sun safety with employee's sun protection practices.
Extraction of costs from parent study ledgers to conduct economic analysis of the SSW intervention. | 9 Months
  Cost information from the SSW parent study project ledgers was extracted for the economic evaluation of the benefits and costs of the intervention.
In-depth manager interview to conduct economic analysis of the SSW intervention. | 9 Months
  An In-depth manger interview was conducted with managers to determine what sun safety items and practices the worksite was doing before and after the program and the costs associated with those practices.
Analysis of employee surveys to compare the impact of workplaces implementing education-only versus education plus policy adoption on employee sun safety practices. | 9 Months
  To compare the actions of intervention employers implementing education, intervention employers implementing education and adopting policy on employee sun safety.

CONTACTS AND LOCATIONS:
Overall Officials: David Buller, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Kaiser Foundation Research Institute, Oakland, California
  - University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No